CLINICAL TRIAL: NCT04136886
Title: Intensity-modulated Radiotherapy Plus Concurrent Chemotherapy Versus Intensity-modulated Radiotherapy Alone In Patients With rT3/T4 Locally Advanced Recurrent Nasopharyngeal Carcinoma: A Phase 3 Multicenter Prospective Randomised Controlled Trial (IMRT)
Brief Title: Concurrent Chemotherapy for Recurrent T3/T4 Nasopharyngeal Carcinoma
Acronym: IMRT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: JiangXi Province Tumor Hospital (Unknown); Fujian Province Tumor Hospital (Other); SiChuan Province Tumor Hospital (Unknown); Hunan Province Tumor Hospital (Other); YuNan Province Tumor Hospital (Unknown); GuiZhou Province Tumor Hospital (Unknown); Hainan Cancer Hospital (Other); Tongji Hospital (Other); Second Affiliated Hospital of Nanchang University (Other); Wuhan University (Other); First Hospital of FoShan City (Unknown)
Responsible Party: Principal Investigator, Fei Han, professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2019-070-01
Record Dates: First submitted 2019-10-22; First posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: concurrent chemotherapy; IMRT; recurrent NPC
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMRT and concurrent cisplatin (Active Comparator): IMRT and concurrent cisplatin to treat T3/T4 locally recurrent NPC patients. Cisplatin 100mg/M2 is to give D1,D22 of IMRT for 2 cycles. IMRT is to give GTV 60Gy in 27 fraction
  Interventions: Drug: Cisplatin; Radiation: IMRT
- IMRT alone (Experimental): IMRT alone to treat T3/T4 locally recurrent NPC patients. IMRT is to give 60Gy in 27 fraction
  Interventions: Radiation: IMRT

INTERVENTIONS:
Drug: Cisplatin — cisplatin is to give from the first Day of radiation therapy D1,D22 Q3W for 2 cycles Radiation: IMRT IMRT is to give 60Gy in 27 fraction
  Arms: IMRT and concurrent cisplatin
Radiation: IMRT — Radiation: IMRT IMRT is to give 60Gy in 27 fraction

SUMMARY:
The purpose of this study is to determine whether concurrent chemotherapy and IMRT is effective in the treatment of locally stage T3/T4 recurrent nasopharyngeal carcinoma patients compared with IMRT alone.

DETAILED DESCRIPTION:
Locally T3/T4 recurrent nasopharyngeal carcinoma (NPC) may be salvaged by intensity modulated-radiotherapy (IMRT), but local control is not good enough and late toxicities is usually severe The aim of this phase III randomized controlled study is to address the efficacy of concurrent chemotherapy (cisplatin) with IMRT to improve local control and lower the occurrence of severe late toxicities compared with IMRT alone for locally T3/T4 recurrent NPC patients.

ELIGIBILITY:
Inclusion Criteria:

* 1.Pathologically or clinically confirmed rT3/T4 locally recurrent nasopharyngeal carcinoma;

  2.No evidence of distant metastasis

  3.More than 1 year from the end of the first course of radiotherapy

  4.Male, or female not in the phase of lactating or pregnancy

  5.ECOG 0-2

  6.Aged 18-70 years old

  7.WBC count ≥4×109/L, neutrophile granulocyte count≥1.5×109/L, PLT count ≥100×109/L, Hb ≥9g/L

  8.Total bilirubin, AST, ALT≤2.0 times of upper normal limits; creatinine ≤1.5 times of upper normal limits

  9.Written informed consort signed

Exclusion Criteria:

1. Only regionally recurrence
2. Evidence of distant metastasis
3. Prior invasive malignancy; noninvasive cancers (For example, carcinoma in situ of the bladder, oral cavity, or cervix are all permissible) are permitted
4. Severe, active co-morbidity
5. Prior anti-tumor treatment after diagnosis of local recurrence
6. MRI was not performed 3 months after the first course of radiotherapy
7. Abnormal function of heart, brain and lungs, etc
8. Lactation or pregnancy
9. Severe nasopharyngeal mucosal necrosis at the diagnosis of local recurrence

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From the beginning the IMRT to 3 year after the end of IMRT

SECONDARY OUTCOMES:
Number of participants with severe acute toxicities as assessed by CTCAE v3.0 | From the beginning of IMRT to 3 months after the end of IMRT
Number of participants with grade 4-5 late adverse events as assessed by RTOG/EORTC Late Radiation Morbidity Scoring Schema | From 3 months after the end of IMRT to 1 year after the end of IMRT

CONTACTS AND LOCATIONS:
Locations (1):
- WangHanYu, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Han F, Zhao C, Huang SM, Lu LX, Huang Y, Deng XW, Mai WY, Teh BS, Butler EB, Lu TX. Long-term outcomes and prognostic factors of re-irradiation for locally recurrent nasopharyngeal carcinoma using intensity-modulated radiotherapy. Clin Oncol (R Coll Radiol). 2012 Oct;24(8):569-76. doi: 10.1016/j.clon.2011.11.010. Epub 2011 Dec 29. PMID 22209574
- [Background] Xiao WW, Huang SM, Han F, Wu SX, Lu LX, Lin CG, Deng XW, Lu TX, Cui NJ, Zhao C. Local control, survival, and late toxicities of locally advanced nasopharyngeal carcinoma treated by simultaneous modulated accelerated radiotherapy combined with cisplatin concurrent chemotherapy: long-term results of a phase 2 study. Cancer. 2011 May 1;117(9):1874-83. doi: 10.1002/cncr.25754. Epub 2010 Nov 16. PMID 21509764
- [Background] Seo Y, Yoo H, Yoo S, Cho C, Yang K, Kim MS, Choi C, Shin Y, Lee D, Lee G. Robotic system-based fractionated stereotactic radiotherapy in locally recurrent nasopharyngeal carcinoma. Radiother Oncol. 2009 Dec;93(3):570-4. doi: 10.1016/j.radonc.2009.10.018. Epub 2009 Nov 16. PMID 19919887
- [Result] Guan Y, Liu S, Wang HY, Guo Y, Xiao WW, Chen CY, Zhao C, Lu TX, Han F. Long-term outcomes of a phase II randomized controlled trial comparing intensity-modulated radiotherapy with or without weekly cisplatin for the treatment of locally recurrent nasopharyngeal carcinoma. Chin J Cancer. 2016 Feb 15;35:20. doi: 10.1186/s40880-016-0081-7. PMID 26879049